CLINICAL TRIAL: NCT01264003
Title: Single Dose Antibiotic Prophylaxis in Lihtenstein Repair for Primary Inguinal Hernias
Brief Title: Antibiotic Prophylaxis in Mesh Repair of Inguinal Hernias
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Diskapi Teaching and Research Hospital (Other)
Responsible Party: 4.Cerrahi Kliniği, Diskapi Teaching and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: DEAH-1002-IHR
Record Dates: First submitted 2010-12-20; First posted 2010-12-21 (Estimated); Last update posted 2010-12-21 (Estimated); Status verified 2008-05

CONDITIONS: Inguinal Hernia
Keywords: inguinal hernia, antibiotic, prophylaxis
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Active Comparator): Antibiotic prohylaxis / Lichtenstein repair
  Interventions: Drug: sefazolin

INTERVENTIONS:
Drug: sefazolin — In prophylaxis

SUMMARY:
Inguinal hernia repairs is clean surgical procedures. However infection may be a concern when prosthetic materials are used. This prospective randomized study has been set to observe if antibiotic prohylaxis is of benefit in mesh repair of inguinal hernias.

DETAILED DESCRIPTION:
There are two group in the study. Control group received no antibiotic prohylaxis, whereas a single dose 1 gr. intravenous cefazoline is given to the patient in prophylaxis arm of the study. 30-days surgical site infection rates and 1 year prosthetic intervention late infection rates are observed and recorded. Side effects of antibiotic used are also recorded.

ELIGIBILITY:
Inclusion Criteria: inguinal hernia repair -

Exclusion Criteria: uncontrolled diabetes mellitus,

-

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2008-05; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Surgical site infection | 30 days postoperatively

SECONDARY OUTCOMES:
Drug side effects | 5 days postoperatively
1-year prosthetic repair surgical site late infection rate | 1 year